CLINICAL TRIAL: NCT00657605
Title: Effects of Human Leptin Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Richard Bookman, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060282; 1R0IDK58851-01 (Other: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK))
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Results first posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Metabolic Syndrome; Diabetes
Keywords: Congenital leptin deficiency; Obesity; Metabolic syndrome; Diabetes
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Diabetes Mellitus | interventions — recombinant methionyl human leptin; metreleptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Recombinant methionyl human leptin (Experimental): Participants with congenital leptin deficiency will receive the Recombinant methionyl human leptin intervention subcutaneously, once a day with a dose of 0.02 to 0.04 mg/kg (adjusted according to weight loss).
  Interventions: Drug: Recombinant methionyl human leptin

INTERVENTIONS:
Drug: Recombinant methionyl human leptin — Recombinant methionyl human leptin, subcutaneous, once a day, 0.02 to 0.04 mg/kg (adjusted according to weight loss), indeterminate duration.
  Other Names: Metreleptin; r-metHuLeptin

SUMMARY:
This study will test the hypothesis that leptin contributes to the regulation of the dynamics of human endocrine function.

DETAILED DESCRIPTION:
The study aims to elucidate the role of leptin in the regulation of human endocrine function approached by a carefully designed, prospective clinical study of the rapidly-sampled dynamics of endocrine rhythms during the course of leptin-replacement treatment in the only three adult individuals identified in the world so far who are leptin-naive due to a functional leptin gene mutation. A study of leptin-naive subjects avoids all confounding factors and pitfalls, because the only bioactive leptin to which they will be exposed is the exogenously administered recombinant protein. Thus, this proposal will permit us to ascertain the endocrine effects of human leptin.

ELIGIBILITY:
Inclusion Criteria:

* Congenital leptin deficiency (these are only 3 adult individuals in the world that have been identified as leptin-naïve thus far).

Exclusion Criteria:

* Pregnant, trying to become pregnant, breast-feeding an infant or sexually active women, not using contraception.
* Subjects with hemoglobin levels below 12 g/dl.
* Subjects whose body contains a ferromagnetic implanted device that might produce a safety hazard during fMRI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2001-06 (Actual); Primary Completion 2010-05-04 (Actual); Study Completion 2010-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Licinio, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Center on Pharmacogenomics, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strobel A, Issad T, Camoin L, Ozata M, Strosberg AD. A leptin missense mutation associated with hypogonadism and morbid obesity. Nat Genet. 1998 Mar;18(3):213-5. doi: 10.1038/ng0398-213. No abstract available. PMID 9500540
- [Result] Baicy K, London ED, Monterosso J, Wong ML, Delibasi T, Sharma A, Licinio J. Leptin replacement alters brain response to food cues in genetically leptin-deficient adults. Proc Natl Acad Sci U S A. 2007 Nov 13;104(46):18276-9. doi: 10.1073/pnas.0706481104. Epub 2007 Nov 6. PMID 17986612
- [Result] Licinio J, Ribeiro L, Busnello JV, Delibasi T, Thakur S, Elashoff RM, Sharma A, Jardack PM, Depaoli AM, Wong ML. Effects of leptin replacement on macro- and micronutrient preferences. Int J Obes (Lond). 2007 Dec;31(12):1859-63. doi: 10.1038/sj.ijo.0803703. Epub 2007 Aug 7. PMID 17684509
- [Result] Licinio J, Milane M, Thakur S, Whelan F, Yildiz BO, Delibasi T, de Miranda PB, Ozata M, Bolu E, Depaoli A, Wong ML. Effects of leptin on intake of specific micro- and macronutrients in a woman with leptin gene deficiency studied off and on leptin at stable body weight. Appetite. 2007 Nov;49(3):594-9. doi: 10.1016/j.appet.2007.03.228. Epub 2007 Apr 6. PMID 17517446
- [Result] Williamson DA, Ravussin E, Wong ML, Wagner A, Dipaoli A, Caglayan S, Ozata M, Martin C, Walden H, Arnett C, Licinio J. Microanalysis of eating behavior of three leptin deficient adults treated with leptin therapy. Appetite. 2005 Aug;45(1):75-80. doi: 10.1016/j.appet.2005.01.002. PMID 15949871
- [Result] Matochik JA, London ED, Yildiz BO, Ozata M, Caglayan S, DePaoli AM, Wong ML, Licinio J. Effect of leptin replacement on brain structure in genetically leptin-deficient adults. J Clin Endocrinol Metab. 2005 May;90(5):2851-4. doi: 10.1210/jc.2004-1979. Epub 2005 Feb 15. PMID 15713712
- [Result] Licinio J, Caglayan S, Ozata M, Yildiz BO, de Miranda PB, O'Kirwan F, Whitby R, Liang L, Cohen P, Bhasin S, Krauss RM, Veldhuis JD, Wagner AJ, DePaoli AM, McCann SM, Wong ML. Phenotypic effects of leptin replacement on morbid obesity, diabetes mellitus, hypogonadism, and behavior in leptin-deficient adults. Proc Natl Acad Sci U S A. 2004 Mar 30;101(13):4531-6. doi: 10.1073/pnas.0308767101. Epub 2004 Mar 9. PMID 15070752
- [Result] Mantzoros CS, Ozata M, Negrao AB, Suchard MA, Ziotopoulou M, Caglayan S, Elashoff RM, Cogswell RJ, Negro P, Liberty V, Wong ML, Veldhuis J, Ozdemir IC, Gold PW, Flier JS, Licinio J. Synchronicity of frequently sampled thyrotropin (TSH) and leptin concentrations in healthy adults and leptin-deficient subjects: evidence for possible partial TSH regulation by leptin in humans. J Clin Endocrinol Metab. 2001 Jul;86(7):3284-91. doi: 10.1210/jcem.86.7.7644. PMID 11443202
- [Result] Ozata M, Ozdemir IC, Licinio J. Human leptin deficiency caused by a missense mutation: multiple endocrine defects, decreased sympathetic tone, and immune system dysfunction indicate new targets for leptin action, greater central than peripheral resistance to the effects of leptin, and spontaneous correction of leptin-mediated defects. J Clin Endocrinol Metab. 1999 Oct;84(10):3686-95. doi: 10.1210/jcem.84.10.5999. PMID 10523015
- [Derived] Paz-Filho G, Wong ML, Licinio J. The procognitive effects of leptin in the brain and their clinical implications. Int J Clin Pract. 2010 Dec;64(13):1808-12. doi: 10.1111/j.1742-1241.2010.02536.x. PMID 21070531
- [Derived] Paz-Filho G, Delibasi T, Erol HK, Wong ML, Licinio J. Congenital leptin deficiency and thyroid function. Thyroid Res. 2009 Nov 4;2(1):11. doi: 10.1186/1756-6614-2-11. PMID 19889232
- [Derived] Paz-Filho G, Esposito K, Hurwitz B, Sharma A, Dong C, Andreev V, Delibasi T, Erol H, Ayala A, Wong ML, Licinio J. Changes in insulin sensitivity during leptin replacement therapy in leptin-deficient patients. Am J Physiol Endocrinol Metab. 2008 Dec;295(6):E1401-8. doi: 10.1152/ajpendo.90450.2008. Epub 2008 Oct 14. PMID 18854428
- [Derived] Andreev VP, Paz-Filho G, Wong ML, Licinio J. Deconvolution of insulin secretion, insulin hepatic extraction post-hepatic delivery rates and sensitivity during 24-hour standardized meals: time course of glucose homeostasis in leptin replacement treatment. Horm Metab Res. 2009 Feb;41(2):142-51. doi: 10.1055/s-0028-1082048. Epub 2008 Aug 22. PMID 18726828

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Recombinant Methionyl Human Leptin
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Recombinant Methionyl Human Leptin
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Time Frame: Baseline, 107 months
Measure: Number; unit: lbs
Arm/Group | Recombinant Methionyl Human Leptin
Number analyzed (Participants) | 3
lbs | NA — Results not reported due to participant confidentiality.

2. Secondary Outcome: Change in Glucose Levels
Time Frame: Baseline, 107 months
Measure: Number; unit: mg/dL
Arm/Group | Recombinant Methionyl Human Leptin
Number analyzed (Participants) | 3
mg/dL | NA — Results not reported due to participant confidentiality.

ADVERSE EVENTS:
Time Frame: 107 months
Description: Adverse Events not reported due to participant confidentiality.
Arm/Group | Recombinant Methionyl Human Leptin
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This is a rare disease population study. To protect participant privacy and maintain confidentiality, results will not be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes